CLINICAL TRIAL: NCT03235466
Title: A Prospective Trial of Behavioral Therapy for Chronic Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Philip Weissbrod, Director, Center for Voice and Swallowing, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181207
Record Dates: First submitted 2017-07-15; First posted 2017-08-01 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of 3 groups: 1) standard voice therapy 2) voice therapy and heart rate variability biofeedback and 3) heart rate variability biofeedback
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Voice Therapy (Active Comparator): (Group 1) will undergo active training in behavioral cough suppression and laryngeal relaxation exercises, but will not receive HRVB. Traditional cough suppression and laryngeal relaxation exercises include pursed lip breathing, swallowing (water, lozenge, gum, ice chips), sustained semi-occluded voicing, discussion and mitigation of triggers, maintaining a cough journal, addressing muscle tension dysphonia if indicated, and developing prophylaxis suppression and laryngeal relaxation based on stimulability. Participants in Group 1 will receive handwritten guidance indicating exercises to practice at home.
  Interventions: Behavioral: Voice Therapy
- Voice Therapy and Heart Rate Variability Biofeedback (Active Comparator): Voice therapy as described in Arm 1. HRVB involves measure respiratory rate, heart rate, body temperature and skin conductance. Participants are guided through reduced breathing rate until a resonant frequency is attained. HRVB breathing simulates resonance between the baroreflex rhythm and respiration based rhythm, increasing heart rate variability and baroreceptor sensitivity. Evidence suggests HRVB improves autonomic regularity. We propose this novel modality to address centrally regulated hypersensitivity that perpetuates coughing.
  Interventions: Behavioral: Voice Therapy and Heart Rate Variability Biofeedback
- Heart Rate Variability Biofeedback (Active Comparator): HRVB as indicated in Arm 2. No instruction will be provided for cough suppression, laryngeal desensitization, voice tasks or hygiene that traditionally reduces cough frequency and severity. This is the experimental arm.
  Interventions: Behavioral: Heart Rate Variability Biofeedback

INTERVENTIONS:
Behavioral: Voice Therapy — See Arm 1 & 2
  Arms: Voice Therapy
Behavioral: Voice Therapy and Heart Rate Variability Biofeedback — See Arm 2 & 3
  Arms: Voice Therapy and Heart Rate Variability Biofeedback
Behavioral: Heart Rate Variability Biofeedback — See Arm 2 & 3
  Arms: Heart Rate Variability Biofeedback

SUMMARY:
This study seeks to explore whether heart rate variability (HRV) biofeedback can be effective in the treatment of chronic cough. Chronic cough has many causes, including asthma, postnasal drip, and gastroesophageal reflux disease (GERD), each with a specific treatment. However, among a subset of cough patients, no clear cause is found despite extensive workup, and traditional treatment methods do not provide relief. Several studies revealed less common causes of chronic cough and disordered breathing such as vagal neuropathy, paradoxical vocal fold motion, and stress. Additional research identified links between the neurological networks that produce the cough reflex and those that maintain normal breathing. HRV biofeedback is a self-regulation technique that uses computer equipment to monitor heart rate and breathing, two key functions of the autonomic nervous system. By using this non-invasive behavioral technique, cough patients can regulate their breathing and autonomic function, potentially leading to improved autonomic balance and a reduction in cough symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 8+ weeks of cough, Fluent English speaker, Have access to an electronic mobile device

Exclusion Criteria:

* On neuromodulator therapy, cardiac arrhythmia, dysphagia, prior HRVB or mindfulness, head and neck surgery of the oropharynx, neck or larynx, lung surgery, pulmonary pathology other than asthma, tourette syndrome, ACE inhibitor use, current or recent smoker.

Added exclusion criteria as of March 2020 - history of COVID+.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Cough reduction | 3 weeks
  Measured by changes in cough severity index and patient recordings

SECONDARY OUTCOMES:
Durability of cough remediation | 8 weeks
  Phone call to patients
Changes in dyspnea | 3 weeks
  Measured by dyspnea index
Change in voice | 3 weeks
  Measured by voice handicap index

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Center for Voice and Swallowing, San Diego, California, United States